CLINICAL TRIAL: NCT02598921
Title: Determining an Accurate and Cost-effective Strategy for Screening for Uterine Cavity Abnormalities in Women Scheduled for IVF
Brief Title: Screening for Uterine Cavity Abnormalities in Women Scheduled for IVF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Khairy Ali, Dr, Assiut University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IVF
Record Dates: First submitted 2015-11-05; First posted 2015-11-06 (Estimated); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Infertility
Keywords: Assisted reproductive technology
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Three dimensional ultrasound (Other): Three dimensional ultrasound evaluated the uterine cavity for cavitary lesions
  Interventions: Radiation: three dimensional ultrasound
- Office hysteroscopy (Other): Office hystrescopy evaluated the uterine cavity for cavitary lesions
  Interventions: Device: Office hysteroscopy

INTERVENTIONS:
Radiation: three dimensional ultrasound
  Arms: Three dimensional ultrasound
Device: Office hysteroscopy
  Arms: Office hysteroscopy

SUMMARY:
Evaluation of the endometrial cavity is an important step in the infertility work-up, particularly if assisted reproductive therapy is planned. The aim is to identify possible endometrial abnormalities that may impair implantation.Undiagnosed endometrial abnormalities are present in 11 to 45% of women scheduled for in vitro fertilization (IVF).Traditionally, two dimensional transvaginal ultrasound (2D TVUS) and hysterosalpingography (HSG) are the basic methods for assessment of the endometrial cavity. However, these imaging modalities have shown high false negative rates among infertile women, a finding that could confine their rule to initial screening rather than definite diagnosis.

Office hysteroscopy (OH) is the gold standard for evaluation of the endometrial cavity. Although the endoscopic approach has been proven to increase pregnancy rate in women who experienced prior implantation failure, evidence on treatment of unsuspected hysteroscopically-diagnosed endometrial lesions, to improve IVF outcome, is still lacking. Nevertheless,clinicians tend to use OH routinely prior to IVF because the psychological and financial burden that infertile couples may experience as a consequence of failed IVF cycle is unjustifiable.Yet, costs and invasiveness of OH counteract its global implementation to all women prior to IVF.

ELIGIBILITY:
Inclusion Criteria:

* History of primary infertility
* Normal uterine cavity on HSG
* Women were selected for IVF therapy.

Exclusion Criteria:

* Women with known diagnosis of uterine abnormality by office hysteroscopy

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2014-07; Primary Completion 2015-08 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Number of patients who have cavitary lesion by three dimensional ultrasound | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt